CLINICAL TRIAL: NCT02643329
Title: Clinical Bioequivalence Study on Two Gliclazide 80mg Tablet Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited (Industry)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BABE-P14-095
Record Dates: First submitted 2015-12-28; First posted 2015-12-31 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
MeSH Terms: interventions — Gliclazide; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BF-Gliclazide Tablet 80mg (Experimental): During the study session, healthy male subjects will be administered a single oral dose of BF-Gliclazide Tablet 80 mg after an overnight fast of approximately 10 hours.
  Interventions: Drug: BF-Gliclazide Tablet 80mg
- Diamicron 80mg Tablet (Active Comparator): During the study session, healthy male subjects will be administered a single oral dose of Diamicron 80 mg Tablet after an overnight fast of approximately 10 hours.
  Interventions: Drug: Diamicron 80mg Tablet

INTERVENTIONS:
Drug: BF-Gliclazide Tablet 80mg — BF-Gliclazide Tablet is a generic product manufactured by Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited
  Other Names: Gliclazide Tablet 80mg
  Arms: BF-Gliclazide Tablet 80mg
Drug: Diamicron 80mg Tablet — Diamicron 80mg Tablet is manufactured by Les Laboratoires Servier Industrie, France
  Other Names: Gliclazide Tablet 80mg
  Arms: Diamicron 80mg Tablet

SUMMARY:
The purpose of the study is to compare the bioavailability of a generic product of gliclazide (Product Name: BF-Gliclazide Tablet 80mg, Manufactured by Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited) with that of reference product (Product Name: Diamicron 80mg Tablet, Manufactured by Les Laboratoires Servier Industrie, France) when administered to healthy volunteers under fasting conditions. The plasma pharmacokinetic data of gliclazide obtained from two formulations will be used to access the interchangeability of the products.

DETAILED DESCRIPTION:
The study design is a single-dose, two-treatment, two-period, two-sequence crossover with a washout period of one to two weeks. During each study session, healthy male subjects will be administered a single oral dose of 80 mg gliclazide (one BF-Gliclazide Tablet 80 mg or one Diamicron 80 mg Tablet) after an overnight fast of approximately 10 hours. 20% glucose will be given orally to each subject at 2 h after drug administration to minimize the risk of hypoglycaemia. Venous blood samples will be collected at pre-dose (0 h) and up to 72 hours post-dose. The plasma concentrations of gliclazide will be determined by a validated assay. The non-compartmental method will be used to analyze the plasma concentration-time data and calculate the main pharmacokinetic parameters such as Cmax, Tmax, AUC0-last, AUC0-inf and T1/2. ANOVA will be conducted on logarithmically transformed Cmax, AUC0-last and AUC0-inf. The two one-sided tests will be used to calculate the 90% confidence intervals for the mean difference in AUC0-last, AUC0-inf and Cmax, and to assess the bioequivalence of the two products.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 18 to 27
* Accessible vein for blood sampling
* High probability for compliance and completion of the study
* No significant abnormalities in general physical examination
* ECG recording within normal limits
* Biochemical and haematological parameters within normal limits
* Subjects must agree to take effective contraceptive methods to prevent his partner from becoming pregnant during the time of first dose of study medication until one week of last dose administration

Exclusion Criteria:

* History of hepatic, renal, biliary, cardiovascular, gastrointestinal, haematological and other chronic and acute diseases within 3 months prior to the study
* Clinically relevant abnormality in physical examination, ECG evaluation, urine test, blood chemistry or haematological test
* Tabacco use in any forms
* Regular consumer of alcohol
* Blood donation within 4 weeks prior to the start of the study
* Use of gliclazide within 4 weeks before the study
* Use of antidiabetic medications within 4 weeks before the study
* Volunteer in any other clinical drug study within 2 months prior to this study
* Hypersensitivity to gliclazide or other drugs in its class
* History of drug abude in any form

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of gliclazide | 72 hours
Area under the plasma concentration versus time curve (AUC) of gliclazide | 72 hours

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) of gliclazide | 72 hours
Elimination half-life (t1/2) of gliclazide | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Vincent HL Lee, Principal Investigator — School of Pharmacy, The Chinese Univesity of Hong Kong; Risa Ozaki, Study Director — Phase 1 Clinical Trial Centre, The Chinese University of Hong Kong; Brian Tomlinson, Study Director — Dept. of Medicine and Therapeutics, The Chinese University of Hong Kong
Locations (1):
- Phase 1 Clinical Trial Centre, The Chinese University of Hong Kong, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Study investigators and his/her study team members, domestic and foreign regulatory agencies, the IRB/EC involved in the study, healthcare providers who provide services to subjects in connection with this study, and laboratories and other individuals and organizations that analyze the subjects' protected health information in connection with this study have access to the data or study.